CLINICAL TRIAL: NCT04267185
Title: Physical Activity Together for MS (PAT-MS): Pilot Study of a Dyadic Rehabilitation Intervention for People with Moderate-to-Severe Multiple Sclerosis Disability and Their Family Caregivers
Brief Title: A Dyadic Approach for Promoting Physical Activity Among People with MS and Their Support Partners
Acronym: PAT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other); Consortium of Multiple Sclerosis Centers (Other); Queen's University (Other)
Responsible Party: Principal Investigator, Lara Pilutti, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190329-01H
Record Dates: First submitted 2020-01-16; First posted 2020-02-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Caregiver; Physical Activity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: This pilot study will use a two-arm, parallel group, single-blinded RCT design that examines the feasibility and preliminary efficacy of a twelve-week physical activity intervention in persons with moderate-to-severe MS disability and their family caregivers compared with a delayed control condition.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be collected objectively by researchers who are blinded to treatment allocation. Researchers who are involved with delivery of the intervention will be aware of treatment allocation, but will not be involved with data collection, entry or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Experimental): PwMS-CG dyads will receive six group telerehabilitation sessions (~60 min each) every other week for a period of 12 weeks. This will be interspersed with brief one-on-one support telephone calls in the weeks that group sessions do not occur. All participants will be taught techniques for monitoring PA behaviour, setting personalized goals to increase PA and reduce sedentary time, and strategies for overcoming challenges to PA participation. Make-up sessions will be offered to those who miss group sessions. The one-on-one support telephone calls will serve to reinforce the information provided during the group sessions, monitor safety and troubleshoot any issues with intervention content.
  Interventions: Behavioral: Physical Activity Together for PwMS and their CGs (PAT-MS)
- Delayed Control (No Intervention): The delayed control group will not receive the intervention during the study period. Participants assigned to the control group will be offered the intervention once the study is completed.

INTERVENTIONS:
Behavioral: Physical Activity Together for PwMS and their CGs (PAT-MS) — A dyadic physical activity intervention approach for PwMS and their family CGs affected by moderate-to-severe MS disability.
  Arms: Immediate Intervention

SUMMARY:
Both people with multiple sclerosis (MS) and their family caregivers experience the impact of this neurodegenerative disease on their health and well-being. The person living with MS and their support partner need to work together as a team to find ways to manage the disease. A physical activity (PA) program that uses a 'dyadic approach' is one possible way of managing the impact of MS. Dyadic programs are unique because they target both people with the disease and their caregivers together to increase their PA levels. This pilot study will deliver a 12-week program using group teleconference and one-on-one support phone calls to teach participants simple methods to change PA patterns in daily life. For example, they will learn how to set personal goals to increase PA and reduce sitting time.

DETAILED DESCRIPTION:
The study is an assessor-blinded pilot randomized controlled trial (RCT) for examining the feasibility and preliminary efficacy of a dyadic PA intervention approach for persons with MS (PwMS) affected by moderate-to-severe disability and their family caregivers (CGs). Dyads who meet the eligibility requirements will undergo the informed consent process and baseline assessment.

Dyads will then be randomized to either an immediate intervention condition or a delayed control condition. Participants in the immediate intervention group will receive six group teleconference sessions, approximately 60 minutes each, every other week for 12 weeks. These sessions will be interspersed with one-on-one support calls in the weeks that group sessions do not occur. Participants will be provided with a manual for their individual use during the intervention. The intervention content will introduce participants to the concepts of shared appraisal and dyadic coping. The benefits of shared participation in PA as a coping strategy to optimize well-being at both the individual and dyadic level will be reinforced and illustrated. All participants will be taught techniques for monitoring PA behaviour, setting personalized goals to increase PA and reduce sedentary time, and strategies for overcoming challenges to PA participation. The one-to-one support calls will serve to reinforce the information provided during the group sessions, monitor safety, and troubleshoot any issues with the intervention content. All participants will undergo the assessment protocol again at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

For persons with MS:

* Physician-confirmed MS diagnosis and stable course of disease modifying therapies over the past 6 months
* Expanded Disability Status Scale (EDSS) score between 6.0 (intermittent or unilateral constant assistance (cane, crutch, brace) required to walk about 100 meters with or without resting) and 6.5 (constant bilateral assistance (canes, crutches, braces) required to walk about 20 meters without resting), based on a Neurostatus-certified assessor examination.
* Relapse-free in the past 30 days
* Support Partner (i.e., relative or close friend) who provides greater than or equal to 1.0 hours per day of unpaid care

Additional inclusion criteria for both persons with MS and caregivers:

* Greater than or equal to 18 years of age
* Currently inactive (i.e., purposeful exercise less than or equal to 2 days/week for 30 minutes)
* Asymptomatic (i.e. no major signs or symptoms of acute or uncontrolled cardiovascular, metabolic, or renal disease) based on the Get Active Questionnaire
* Ability to communicate in English

Exclusion Criteria for both persons with MS and caregivers:

* diagnosis of other neurological condition(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Safety of the PAT-MS intervention | Assessed weekly through study completion at 12 weeks
  Safety will be recorded via reporting of adverse events (AEs) during testing sessions and one-on-one support calls. AEs will be defined as any unfavorable change in health that occurs in both PwMS and CGs during the trial period, e.g. injuries, relapses, falls and symptomatic changes. Each AE will be rated based on severity, expectedness, and potential relation to study participation using the Common Terminology for Adverse Events (CTCAE) classification scheme. AEs will be reported as the overall rate, severity, and characteristics of the events.
Feasibility: Participant recruitment rate | Recorded through the 6-month recruitment period
  We will use phone call and electronic mail recruitment and record all contact with potential participants and refusal reasons.
Feasibility: Participant compliance rate | Recorded weekly through study completion at 12 weeks
  Will be assessed by recording the number of practice activities, group teleconference sessions, and one-on-one phone calls completed by participants.
Feasibility: Participant attrition rate | Will be assessed at T2 (12 Weeks)
  Will be assessed as the percentage of the sample who drop out of the study.
Feasibility: Monetary cost of research | Recorded from study initiation to completion, approximately 2 years
  We will establish and record all monetary costs for the study.
Feasibility: Staff time | Recorded weekly through study completion at 12 weeks
  We will document all preparation, call time, attempted call time and report-taking time for each participant during the intervention.
Feasibility: Research ethics procedures | Recorded from study initiation to completion, approximately 2 years
  We will document communications between the research ethics board and staff, and time from submission of research ethics application to approval.
Feasibility: Data collection at T1 | Will be assessed at T1 (Baseline)
  We will check for data completeness, and record time to collect, enter and check data in a database
Feasibility: Data collection at T2 | Will be assessed at T2 (12 Weeks)
  We will check for data completeness, and record time to collect, enter and check data in a database
Change in Self-Reported Physical Activity - Primary Efficacy Outcome | Change in Self-reported PA (total PA minutes) between T1 (Baseline) and T2 (12 Weeks)
  Change in Self-reported physical activity (PA) level of PwMS and CGs will be assessed using the Godin Leisure-Time Exercise Questionnaire (GLTEQ). The GLTEQ has been demonstrated to be a reliable and valid primary outcome for measuring change in PA in response to a behavioural intervention.

SECONDARY OUTCOMES:
Change in Accelerometer-measured Physical Activity - steps/day | Change in accelerometer-measured steps/day between T1 (Baseline) and T2 (12 Weeks).
  Accelerometer-measured PA will be assessed as steps/day in both PwMS and CGs. At each assessment session, both PwMS and CGs will be provided with an Actigraph Activity monitor (accelerometer) to take home, along with a logbook to record the time periods in which the accelerometer was worn. Participants will be instructed to wear the accelerometer during all waking hours, except while engaging in water activities.
Change in Accelerometer-measured Physical Activity - minutes of PA | Change in accelerometer-measured minutes of PA between T1 (Baseline) and T2 (12 Weeks).
  Accelerometer-measured PA will be assessed as minutes spent in sedentary behaviour, light activity, and moderate-to-vigorous activity in both PwMS and CGs. At each assessment session, both PwMS and CGs will be provided with an Actigraph Activity monitor (accelerometer) to take home, along with a logbook to record the time periods in which the accelerometer was worn. Participants will be instructed to wear the accelerometer during all waking hours, except while engaging in water activities.
Change in Walking Speed | Change in walking speed between T1 (Baseline) and T2 (12 Weeks).
  Walking speed will be assessed in PwMS using the timed 25-foot walk (T25FW) test. The T25FW test will involve participants walking as quickly and safely as possible across a 25-foot distance. Participants will be asked to complete two walking trials and the average walking speed of the two trials will be reported in meters/second.
Change in Walking Endurance | Change in Walking endurance between T1 (Baseline) and T2 (12 Weeks)
  Walking endurance will be assessed in PwMS using the 2-minute walk (2MW) test. The 2MW test involves participants walking as fast and as far as possible in an accessible hallway for 2 minutes. Participants will complete one walking trial.
Change in Agility | Change in Agility between T1 (Baseline) and T2 (12 Weeks).
  Agility will be assessed in PwMS using the Timed Up-and-Go (TUG) test. The TUG test involves participants rising from a chair, walking 3 meters, turning around, and then walking back to the chair and returning to the seated position. Participants will complete two trials of the TUG test. The time taken in seconds for each trial will be recorded.
Change in Physical Functional Limitations and Disability | Change in Physical functional limitations and disability between T1 (Baseline) and T2 (12 Weeks).
  Physical functional limitations and disability will be assessed in PwMS using the abbreviated Late-Life Function and Disability Instrument (LLFDI) questionnaire. The LLFDI contains fifteen items within 3 subscales: basic lower extremity function, advanced lower extremity function, and upper extremity function. A composite score is generated by summing all three subscale scores. Higher scores indicate fewer functional limitations.
Change in MS Self-Efficacy | Change in MS self-efficacy between T1 (Baseline) and T2 (12 Weeks).
  Self-efficacy will be assessed in PwMS using the MS Self-Efficacy (MSSE) Scale. The questionnaire is an 18-item scale divided into 2 subscales: function and control. The items assess how confident individuals feel that they can achieve a specific function or control various aspects of their MS. Scores are totaled on each subscale and a total MSSE is obtained. Higher scores are associated with higher degrees of certainty.
Change in Quality of Life in PwMS | Change in Quality of life in PwMS between T1 (Baseline) and T2 (12 Weeks).
  Quality of life will be assessed in PwMS using the MS Impact Scale-29 (MSIS-29). The MSIS-29 questionnaire is a measure of physical and psychological health-related quality of life. Higher scores indicate a greater physical and psychological impact of MS on daily activities.
Change in Dyadic Relationship Quality | Change in Dyadic relationship quality between T1 (Baseline) and T2 (12 Weeks)
  Dyadic relationship quality will be assessed both in PwMS and CGs using the Short-form Dyadic Adjustment Scale. The questionnaire consists of 7 items rated on a 5-point Likert scale. Higher scores indicate greater relationship quality.
Change in Perceptions of Social Support | Change in perceptions of social support between T1 (Baseline) and T2 (12 Weeks).
  Perceptions of social support will be assessed in both PwMS and CGs using the Interpersonal Support Evaluation List-12 (ISEL-12). This 12-item questionnaire is designed to measure 3 subscales (appraisal, belonging, and tangible) of perceived social support. Each item is rated on a 4-point scale.
Change in Resilience | Change in Resilience between T1 (Baseline) and T2 (12 Weeks).
  Resilience will be assessed in both PwMS and CGs using the Conner-Davidson Resilience Scale (CD-RISC-10). The questionnaire evaluates perceived ability to deal with stressful and challenging situations and to overcome obstacles.
Change in Coping | Change in Coping in CGs between T1 (Baseline) and T2 (12 Weeks).
  Coping will be assessed in CGs using the Coping with MS Caregiving Inventory (CMSCI). The questionnaire is a measure of 34 coping strategies specific to MS caregiving. Respondents indicate on a 4-point scale how often they have used each of the coping strategies in dealing with caregiving in general in the past month.
Change in Quality of Life in Caregivers | Change in Quality of life in CGs between T1 (Baseline) and T2 (12 Weeks).
  Quality of life in CGs will be assessed using the Caregiver Quality of Life in MS scale (CAREQOL-MS). The questionnaire is a measure of caregiver health-related quality of life. The scale consists of 24 items comprising the four subscales of physical stress/global health, social integration, emotion, and the need for assistance/emotional reactions. Items are scored using a 5-point Likert-type scale with higher scores reflecting worse quality of life.

OTHER OUTCOMES:
Satisfaction Survey | T2 (12 Weeks)
  All participants in the Immediate Intervention group will be asked to complete a 10-item satisfaction survey developed for this study to asses their experience of study involvement. Items are scored on a 5-point Likert scale with higher scores reflecting higher satisfaction.
Experiential Aspects of Participation | T2 (12 Weeks)
  Experiential aspects of physical activity participation will be assessed in participants in the Immediate Intervention group using the Measure of Experiential Aspects of Participation (MeEAP). The scale consists of 12 items comprising the six subscales of autonomy, belongingness, mastery, challenge, engagement, and meaning. Items are scored using a 7-point Likert-type scale with higher scores reflecting higher quality of participation.
Semi-structured Qualitative Interview | T2 (12 Weeks)
  PwMS and their CGs who complete the 12-week physical activity intervention will be asked to participate in an optional telephone qualitative interview to further explore their experiences of participating in the intervention, perceptions of benefits, and suggestions for improvement. Telephone interviews will involve participants chosen at random from those who indicated that they would be willing to be interviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pilutti, PhD, Principal Investigator — University of Ottawa; Mark Freedman, MD, Principal Investigator — The Ottawa Hospital/Ottawa Hospital Research Institute
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fakolade A, Lamarre J, Latimer-Cheung A, Parsons T, Morrow SA, Finlayson M. Understanding leisure-time physical activity: Voices of people with MS who have moderate-to-severe disability and their family caregivers. Health Expect. 2018 Feb;21(1):181-191. doi: 10.1111/hex.12600. Epub 2017 Jul 19. PMID 28722772
- [Background] Fakolade A, Latimer-Cheung A, Parsons T, Finlayson M. A concerns report survey of physical activity support needs of people with moderate-to-severe MS disability and family caregivers. Disabil Rehabil. 2019 Dec;41(24):2888-2899. doi: 10.1080/09638288.2018.1479781. Epub 2018 Jun 29. PMID 29958014
- [Background] Fakolade A, Finlayson M, Parsons T, Latimer-Cheung A. Correlating the Physical Activity Patterns of People with Moderate to Severe Multiple Sclerosis Disability and Their Family Caregivers. Physiother Can. 2018 Fall;70(4):373-381. doi: 10.3138/ptc.2017-36.ep. PMID 30745723
- [Derived] Fakolade A, Awadia Z, Cardwell K, McKenna O, Venasse M, Hume T, Ludgate J, Freedman MS, Finlayson M, Latimer-Cheung AE, Pilutti LA. Physical Activity Together for Multiple Sclerosis (PAT-MS): A randomized controlled feasibility trial of a dyadic behaviour change intervention. Contemp Clin Trials Commun. 2023 Oct 16;36:101222. doi: 10.1016/j.conctc.2023.101222. eCollection 2023 Dec. PMID 37928934
- [Derived] Fakolade A, Cameron J, McKenna O, Finlayson ML, Freedman MS, Latimer-Cheung AE, Pilutti LA. Physical Activity Together for People With Multiple Sclerosis and Their Care Partners: Protocol for a Feasibility Randomized Controlled Trial of a Dyadic Intervention. JMIR Res Protoc. 2021 Jun 1;10(6):e18410. doi: 10.2196/18410. PMID 34061040